CLINICAL TRIAL: NCT00436215
Title: A Phase II Study of Sorafenib and Bevacizumab in Epithelial Ovarian, Fallopian, and Peritoneal Cancer
Brief Title: Sorafenib and Bevacizumab to Treat Ovarian, Fallopian and Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christina Annunziata, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070058; 07-C-0058
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2015-03-26 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Ovarian Neoplasm; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: Sorafenib; Ovarian Cancer; Fallopian Cancer; Bevacizumab; Peritoneal Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Bevacizumab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BAY 43-9006 + Bevacizumab (Experimental): BAY 43-9006 (sorafenib) + Bevacizumab
  Interventions: Drug: Bevacizumab; Drug: BAY 43-9006

INTERVENTIONS:
Drug: Bevacizumab — bevacizumab 5 mg/kg intravenous (IV) every two weeks
  Other Names: Avastin
Drug: BAY 43-9006 — BAY 43-9006 200 mg po (by mouth) twice daily 5 out of 7 days each week (Mon-Fri)
  Other Names: sorafenib

SUMMARY:
Background:

* Sorafenib and bevacizumab are anti-cancer drugs that work by targeting the blood vessels that allow tumors to grow. Using the two drugs together may more effectively block the formation of blood vessels that feed tumors.
* Sorafenib and bevacizumab both are approved by the Food and Drug Administration for use in other cancers but have not ovarian cancer. In a preliminary trial of this drug combination, however, tumors in 6 of 14 patients with ovarian cancer shrank.

Objectives:

* To determine the safety and activity of the combination of sorafenib and bevacizumab for treating patients with ovarian, fallopian and peritoneal cancer.
* To determine how sorafenib and bevacizumab may affect the cancer by measuring amounts of different proteins in small biopsy samples of tumor taken before starting treatment and after 6 weeks.

Eligibility:

* Females 18 years of age and older with ovarian, fallopian, or peritoneal cancer whose disease has not responded to standard treatment or for which no standard treatment is available.
* Patients must have not been previously treated with bevacizumab or must have had their disease worsen while taking bevacizumab-based therapy.

Design:

* Patients take 200 mg of sorafenib by mouth twice a day Monday through Friday each week and 5 mg/kg of bevacizumab through a vein every 2 weeks.
* Tumor biopsies and imaging scans (magnetic resonance imaging (MRI) and positron emission tomography (PET) are done before treatment, 3 days after beginning treatment, and 6 weeks into therapy.
* Computed tomography (CT) or other imaging tests are done every 8 weeks to evaluate response to treatment.
* History, physical examinations, blood and urine tests are done periodically during treatment for health checks and research purposes.
* About 74 patients are to be enrolled in the trial.

DETAILED DESCRIPTION:
Background:

Sorafenib is an inhibitor of wild-type and mutant proto-oncogene BRaf (B-Raf) and proto-oncogene c-Raf (c-Raf) kinase isoforms in vitro, but it also inhibits mitogen-activated protein kinase (p38), proto-oncogene c-kit (c-kit), vascular endothelial growth factor receptor 2 (VEGFR-2) and platelet-derived growth factor (PDGFR)-Beta affecting tumor growth as well as possibly promoting apoptosis by events downstream of c-Raf.

Bevacizumab is a humanized immunoglobulin G 1 (IgG1) monoclonal antibody (MAb) that binds all biologically active isoforms of human vascular endothelial growth factor (vascular endothelial growth factor (VEGF), or VEGF-A) with high affinity (kd = 1.1nM).

Phase I trial of sorafenib and bevacizumab administered concurrently showed activity of the combination in patients with refractory ovarian cancer.

Objectives:

Determine the activity and tolerability of the combination bevacizumab and sorafenib in patients with refractory or recurrent epithelial ovarian, fallopian, or peritoneal cancer in patients who are bevacizumab-naive or bevacizumab-resistant.

Eligibility:

Adults with histologically documented refractory or recurrent epithelial ovarian, fallopian, or peritoneal cancer.

Patients must be off prior chemotherapy, radiation therapy, hormonal therapy, or biological therapy for at least 4 weeks.

Patients must have an Eastern Cooperative Oncology Group (ECOG) of 1 or less.

Patients must have disease that is amenable to biopsy.

Patients must have not been previously treated with bevacizumab or must have progressed on prior bevacizumab-based therapy.

Design:

Patients will be stratified on entrance to the trial based on their previous exposure to bevacizumab to either strata A (bevacizumab-naive patients) or strata B (patients previously treated with bevacizumab).

Patients will receive oral sorafenib 200 mg twice daily 5 out of 7 days each week and intravenous bevacizumab 5 mg/kg every two weeks.

Tumor biopsies will be obtained from patients before treatment and six weeks into therapy. Dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) and fludeoxyglucose 18F-positron emission tomography (FDG-PET) will be obtained from patients before treatment, on day 3 of treatment, and six weeks into therapy.

Patients will be evaluated for response every 8 weeks using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

Approximately 74 patients will be needed to achieve the objectives of the trial.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Histopathologically documented recurrent/refractory epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer from a previous biopsy verified by the Laboratory of Pathology, National Cancer Institute (NCI).

-Recurrent/refractory disease defined as progression within 6 months of upfront platinum-containing therapy or progression after subsequent therapy in previously relapsed patients.

Disease amenable to percutaneous or skin biopsy as determined by an associate investigator and a member of the interventional team.

Patient willingness to have biopsies performed.

Measurable disease defined as tumor greater than or equal to 1 cm.

Age greater than or equal to 18 years.

Life expectancy of more than 3 months.

Performance status of 0 to 1 according to the Eastern Cooperative Oncology Group (ECOG) criteria.

Adequate organ function as defined below:

Laboratory Test Required value

* Leukocytes greater than or equal to 3,000/ microliter
* Absolute neutrophil count greater than or equal to 1,200/ microliter
* Platelets greater than or equal to 100,000/ microliter
* Total bilirubin less than or equal to 1.5 times the institutional upper limits of normal
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 times the institutional upper limit of normal
* Creatinine less than or equal to 1.5 mg/dL

OR

* Creatinine clearance greater than or equal to 45 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.
* Activated partial thromboplastin time (PTT) less than 1.5 times the institutional upper limits of normal
* Prothrombin Time (PT)/ International normalized ratio (INR) less than 1.5 times the institutional upper limits of normal
* Amylase and Lipase Less than institutional upper limits of normal

Patients must have a urine protein/creatinine ratio (UPC) less than 1.0 for enrollment.

No surgery, radiation therapy, chemotherapy, immunotherapy, biotherapy, or hormonal therapy (exception raloxifene for bone health) within four weeks (6 weeks for mitomycin C, carboplatin, or nitrosoureas);

No metabolically active complimentary or alternative therapy for at least 1 week, defined as any ingested or administered chemical substances including herbal medications, but not including acupuncture, hypnosis, meditation, or other non-chemical treatments.

No monoclonal antibody therapy for at least 6 weeks.

Patients must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be less than or equal to grade 1 (as defined by Common Terminology Criteria for Adverse Events (CTCAE v3) or returned to baseline. Peripheral neuropathy less than or equal to grade 2 will be allowed as this patient population has universally been treated with platinum-based chemotherapy with residual neuropathy being a common occurrence.

No other invasive malignancies within the past two years (with the exception of non-melanoma skin cancers, non-invasive bladder cancer, stage I endometrial cancer or cervical cancer synchronous to the ovarian cancer diagnosis and cured by surgical resection).

Ability to understand and sign an informed consent form.

Patients who require hematopoietic growth factor support (e.g. epogen, darbepoetin), Non-steroidal anti-inflammatory drugs (NSAIDs), and other maintenance medications prior to study entry will be allowed to continue their supportive therapies.

Ability to tolerate orally administered medications.

Contraception is not a consideration as these patients have all had surgical removal of their reproductive organs. Pregnant women are excluded from this study because BAY 43-9006 and bevacizumab are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with BAY 43-9006 and/or bevacizumab, breastfeeding should be discontinued if the mother is treated with BAY 43-9006 and/or bevacizumab.

There is no limit on the number of prior regimens with which a patient has been treated.

Patients who have been treated with bevacizumab previously are eligible for the trial if they have progressed while on bevacizumab-based therapy.

-Disease progression on bevacizumab therapy will be defined as documented increase in disease based on imaging while the patient is receiving bevacizumab or within three months of their last dose of bevacizumab.

Patients must be at least 6 weeks from their last dose of bevacizumab prior to being enrolled on study.

Patients who have a healed fistula greater than 28 days prior to enrollment are eligible (refer to section 3.2.15 for patients who have had prior bevacizumab)

EXCLUSION CRITERIA:

Serious non-healing wounds (including wounds healing by secondary intention), acute or non-healing ulcers, or bone fractures within 3 months of enrollment.

Moderate or massive hemoptysis or surgery within 28 days of enrollment.

Ongoing treatment with any other investigational agents.

Brain metastases

* Patients with central nervous system (CNS) metastases within the past 2 years are ineligible. Patients who have had CNS disease curatively treated and without recurrence for 2 years may be eligible. but any CNS disease that has not undergone curative therapy with radiation, gamma knife, and/or surgical therapy are ineligible.
* CNS imaging will not be mandated for all patients. However, if there is clinical suspicion of CNS involvement, a contrast computed tomography (CT) or magnetic resonance imaging (MRI) of the brain will be required.
* Patients with CNS metastases may not be on steroids for the purpose of CNS disease or edema control.
* Patients with CNS disease must be on an anti-seizure medication and that medication cannot be a CYPP4503A modulating agent.

Thrombotic or embolic events within the past 6 months such as a cerebrovascular accident (including transient ischemic attacks), pulmonary embolism, unstable angina, or myocardial infarction. Fully treated deep vein thrombosis no longer requiring anticoagulation will be allowed.

Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (American Heart Association (AHA) Class II or worse), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

-Patients with evidence of active infection will become eligible for reconsideration 7 days after completing antibiotic therapy.

Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with sorafenib, bevacizumab, and/or the combination.

Hypertension defined as systolic blood pressure greater than 150 mmHg or diastolic pressure greater than 90 mmHg despite optimal medical management.

Therapeutic anticoagulation with coumadin, heparins, or heparinoids.

Evidence of a bleeding diathesis.

History of high grade varices or arteriovenous malformations.

Patients previously treated with sorafenib will not be eligible for this trial.

Fistula or bowel obstruction or perforation in the 28 days prior to enrollment.

Patients must not be taking the cytochrome p450 (CYP450) enzyme-inducing drugs phenytoin, carbamazepine, phenobarbital, St. John's wort, or rifampin.

For patients who have been previously treated with bevacizumab, any severe toxicity associated with bevacizumab while the patient was being treated with the agent will make the patient ineligible for the trial. This includes bevacizumab-induced hypertensive crisis, arterial thromboembolic events (including cardiac ischemia or cerebrovascular ischemia or other arterial thrombosis), nephrotic syndrome, gastrointestinal perforation, serious hemorrhage, and fistulas (unless the fistula completely resolved while the patient was still on bevacizumab or it has been surgically corrected).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Histopathologically documented recurrent/refractory epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer from a previous biopsy verified by the Laboratory of Pathology, National Cancer Institute (NCI).
Enrollment: 55 (Actual)
Dates: Start 2006-12-12 (Actual); Primary Completion 2014-06-26 (Actual); Study Completion 2014-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Annunziata, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singer G, Oldt R 3rd, Cohen Y, Wang BG, Sidransky D, Kurman RJ, Shih IeM. Mutations in BRAF and KRAS characterize the development of low-grade ovarian serous carcinoma. J Natl Cancer Inst. 2003 Mar 19;95(6):484-6. doi: 10.1093/jnci/95.6.484. PMID 12644542
- [Background] Cohen Y, Xing M, Mambo E, Guo Z, Wu G, Trink B, Beller U, Westra WH, Ladenson PW, Sidransky D. BRAF mutation in papillary thyroid carcinoma. J Natl Cancer Inst. 2003 Apr 16;95(8):625-7. doi: 10.1093/jnci/95.8.625. PMID 12697856
- [Background] Pollock PM, Meltzer PS. A genome-based strategy uncovers frequent BRAF mutations in melanoma. Cancer Cell. 2002 Jul;2(1):5-7. doi: 10.1016/s1535-6108(02)00089-2. PMID 12150818
- [Result] Lee JM, Annunziata CM, Hays JL, Cao L, Choyke P, Yu M, An D, Turkbey IB, Minasian LM, Steinberg SM, Chen H, Wright J, Kohn EC. Phase II trial of bevacizumab and sorafenib in recurrent ovarian cancer patients with or without prior-bevacizumab treatment. Gynecol Oncol. 2020 Oct;159(1):88-94. doi: 10.1016/j.ygyno.2020.07.031. Epub 2020 Aug 1. PMID 32747013
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-C-0058.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BAY 43-9006 + Bevacizumab
Started | 55
Completed | 51
Not Completed | 4
Not completed — Refused further treatment | 3
Not completed — Small bowel obstruction | 1

BASELINE CHARACTERISTICS:
Arm/Group | BAY 43-9006 + Bevacizumab
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.37 (12.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 51
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rate.
Description: Clinical response rate is defined as the percentage of participants with a complete response (CR) or partial response (PR) per the Response Evaluation Criteria in Solid Tumors (RECIST). CR is disappearance of all target lesions. PR is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive disease (PD) is a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease (SD) is neither sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started lasting at least 6 months.
Time Frame: patients were followed for a median of 18 weeks (range 1-116 weeks)
Population: Seven patients were not evaluable for response assessment.
Measure: Number; unit: percentage of participants
Arm/Group | BAY 43-9006 + Bevacizumab
Number analyzed (Participants) | 48
percentage of participants
  Complete Response | 0
  Partial Response | 19
  Progressive Disease | 21
  Stable Disease | 60

2. Secondary Outcome: Progression-free Survival
Description: Progression free survival is defined by the number of weeks between the first day of treatment and the date of cancer progression.
Time Frame: up to 28 months
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | BAY 43-9006 + Bevacizumab
Number analyzed (Participants) | 55
Weeks | 26 (24)

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: up to 28 months
Measure: Count of Participants; unit: Participants
Arm/Group | BAY 43-9006 + Bevacizumab
Number analyzed (Participants) | 55
Participants | 54

ADVERSE EVENTS:
Time Frame: up to 28 months
Arm/Group | BAY 43-9006 + Bevacizumab
All-Cause Mortality (participants affected / at risk) | 1/55
Serious Adverse Events (participants affected / at risk) | 25/55
Other Adverse Events (participants affected / at risk) | 54/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAY 43-9006 + Bevacizumab (N=55)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Allergic reaction (Immune system disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Cecal infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hepatobiliary disorders - Other, specify (bile duct obstruction) (Hepatobiliary disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Obstruction gastric (Gastrointestinal disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 7 (7)
Thromboembolic event (Vascular disorders) | 4 (5)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAY 43-9006 + Bevacizumab (N=55)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 14 (16)
Activated partial thromboplastin time prolonged (Investigations) | 20 (38)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 30 (58)
Alkaline phosphatase increased (Investigations) | 23 (46)
Allergic reaction (Immune system disorders) | 2 (2)
Allergic rhinitis (Immune system disorders) | 7 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anal mucositis (Gastrointestinal disorders) | 1 (1)
Anal pain (Gastrointestinal disorders) | 2 (2)
Anaphylaxis (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 13 (21)
Anorectal infection (Infections and infestations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 17 (22)
Anxiety (Psychiatric disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 38 (65)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10)
Blood bilirubin increased (Investigations) | 10 (14)
Blurred vision (Eye disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1)
CPK increased (Investigations) | 3 (4)
Cataract (Eye disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Chills (General disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Creatinine increased (Investigations) | 10 (22)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Depression (Psychiatric disorders) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 17 (35)
Dizziness (Nervous system disorders) | 6 (6)
Dry eye (Eye disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 10 (10)
Dyspepsia (Gastrointestinal disorders) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 (19)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Eye pain (General disorders) | 2 (2)
Fatigue (General disorders) | 26 (28)
Fever (General disorders) | 6 (8)
Flashing lights (Eye disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (early satiety) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (gastroenteritis) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 22 (30)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 3 (4)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 5 (5)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Hot flashes (Vascular disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 11 (17)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 12 (15)
Hypertension (Vascular disorders) | 30 (49)
Hyperthyroidism (Endocrine disorders) | 9 (9)
Hyperuricemia (Metabolism and nutrition disorders) | 7 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 41 (85)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 6 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 23 (50)
Hyponatremia (Metabolism and nutrition disorders) | 31 (75)
Hypoparathyroidism (Endocrine disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 11 (15)
Hypotension (Vascular disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 4 (4)
Infections and infestations - Other, specify (bronchitis) (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (oral candidasis/thrush) (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (pyuria) (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (unknown ANC) (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — viral syndrome (fever), normal ANC
Infections and infestations - Other, specify (Infections and infestations) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (6)
Investigations - Other, specify (Investigations) | 2 (2)
Lethargy (Nervous system disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1)
Lipase increased (Investigations) | 6 (13)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 26 (69)
Memory impairment (Nervous system disorders) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 35 (59)
Musculoskeletal and connective tissue disorder - Other, specify (cramps) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (muscle cramping) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — muscle spasm (back) intermittent
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 18 (21)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (2)
Neutrophil count decreased (Investigations) | 3 (4)
Non-cardiac chest pain (General disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (3)
Pain (General disorders) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (11)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 47 (104)
Paresthesia (Nervous system disorders) | 1 (3)
Pelvic pain (Reproductive system and breast disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Phlebitis infective (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 19 (27)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Proctitis (Gastrointestinal disorders) | 3 (4)
Proteinuria (Renal and urinary disorders) | 13 (18)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (11)
Rash acneiform (Skin and subcutaneous tissue disorders) | 12 (15)
Rash maculo-papular (Gastrointestinal disorders) | 9 (10)
Rectal hemorrhage (Gastrointestinal disorders) | 3 (3)
Rectal pain (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (dysuria) (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (high blood urea nitrogen) (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (WBC in urine) (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Renal hemorrhage (Renal and urinary disorders) | 1 (2)
Rhinitis infective (Infections and infestations) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 2 (3)
Serum amylase increased (Investigations) | 6 (12)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Sinusitis (Infections and infestations) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — blisters, heel
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2) — brittle hair
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — keratosis pilaris
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — perianal rash (HSV)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2)
Skin infection (Infections and infestations) | 4 (4)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 11 (12)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 8 (9)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 3 (3)
Vaginal infection (Infections and infestations) | 3 (3)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Vomiting (Gastrointestinal disorders) | 11 (16)
Weight gain (Investigations) | 2 (3)
Weight loss (Investigations) | 29 (44)
White blood cell decreased (Investigations) | 10 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT00436215/Prot_SAP_000.pdf
  • Informed Consent Form (2014-05-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT00436215/ICF_001.pdf